CLINICAL TRIAL: NCT00252811
Title: A Phase II, Randomised, Double-Blind, Placebocontrolled Study To Investigate The Effects Of ZD1839 (IRESSA™) On Cell Proliferation In Oestrogen And Progesterone Receptor Negative Breast Cancer Prior To Surgery
Brief Title: A Study of ZD1839 Effects on Cell Proliferation in Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0509; D7913C00509 (Other: AZ IMPACT)
Record Dates: First submitted 2005-11-01; First posted 2005-11-15 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib

SUMMARY:
This is a Phase II, randomised, double-blind, placebo-controlled study. Subjects with histologically-confirmed oestrogen receptor negative (ER-), progesterone receptor negative (PgR-) primary breast cancer breast cancer will be randomly assigned in a 2:1 ratio to receive ZD1839 250 mg once daily or matching placebo for a total period of 5 weeks. Surgical intervention will take place after 4 weeks (on Day 29) and treatment will continue for 1 week after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed ER- and PgR- primary breast cancer
* Stage T .5 cm, N0-1, M0
* No previous treatment for breast cancer

Exclusion Criteria:

* ALT or AST greater than 2.5 times the ULRR
* Metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-02

PRIMARY OUTCOMES:
Estimate the effect of ZD1839 compared with placebo on the change in tumour cell proliferation in patients who have completely ER negative & PgR negative breast cancer
Aassessment of biomarker Ki-67 in breast cancer tissue at baseline by core biopsy and after 4 weeks on the surgical specimen

SECONDARY OUTCOMES:
To assess the effect of 4 weeks of ZD1839 on the change in tumour size as assessed by ultrasounds.
To correlate the expression of tissue biomarkers (HER family and epidermal growth factor [EGF] related pathways) in the baseline biopsy sample and in the surgical (endpoint) specimen with the anti-proliferative effect of ZD1839.
To determine the effect of ZD1839 on HER-2 phosphorylation and other biomarkers in the surgical (endpoint) specimens when compared with the baseline biopsies
To assess the effect of ZD1839 on apoptosis as assessed by TUNEL in the surgical (endpoint) specimens when compared with the baseline biopsies
To determine plasma trough concentrations of ZD1839 and correlate these with molecular biomarkers detected in breast cancer tissue.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Italy Medical Director, MD, Study Director — AstraZeneca; A Decensi, MD, Principal Investigator — Istituto Europeo di Oncologia di Milano
Locations (1):
- Research Site, Milan, Italy